CLINICAL TRIAL: NCT05832502
Title: A Placebo Controlled Clinical Trial Investigating the Safety and Immunogenicity of GBS6 in Pregnant Women With and Without Human Immunodeficiency Virus (HIV) Infection and Their Infants
Brief Title: Clinical Trial Investigating the Safety and Immunogenicity of GBS6 in Pregnant Women With and Without HIV (PREPARE)
Acronym: PREPARE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Collaborators: MU-JHU CARE (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020.0317
Record Dates: First submitted 2023-02-20; First posted 2023-04-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-11

CONDITIONS: Group B Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (saline) in HIV-uninfected pregnant woman (Placebo Comparator): Placebo (saline control) administered intramuscularly by injecting 0.5 mL into the deltoid muscle
  Interventions: Drug: Placebo
- GBS6 in HIV-uninfected pregnant woman (Active Comparator): GBS6 administered intramuscularly by injecting 0.5 mL into the deltoid muscle
  Interventions: Drug: GBS6
- Placebo (saline) in HIV-infected pregnant woman (Placebo Comparator): Placebo (saline control) administered intramuscularly by injecting 0.5 mL into the deltoid muscle
  Interventions: Drug: Placebo
- GBS6 in HIV-infected pregnant woman (Active Comparator): GBS6 administered intramuscularly by injecting 0.5 mL into the deltoid muscle
  Interventions: Drug: GBS6

INTERVENTIONS:
Drug: GBS6 — The investigational products are GBS6 and placebo (saline control). The GBS6 dose will be GBS6 20mcg without AlPO4 (equivalent to 240 mcg/mL) 0.5mL dose or 20 mcg CPS/serotype).
  Other Names: Hexavalent anti capsular polysaccharide (CPS) / cross reactive material 197 glycoconjugate
  Arms: GBS6 in HIV-infected pregnant woman; GBS6 in HIV-uninfected pregnant woman
Drug: Placebo — Placebo (saline control) administered intramuscularly by injecting 0.5 mL into the deltoid muscle
  Arms: Placebo (saline) in HIV-infected pregnant woman; Placebo (saline) in HIV-uninfected pregnant woman

SUMMARY:
A placebo controlled clinical trial investigating the safety and immunogenicity of GBS6 in pregnant women with and without human immunodeficiency virus (HIV) infection and their infants

DETAILED DESCRIPTION:
This Phase 2, randomised, placebo controlled, double blinded study will be the first evaluation of the investigational GBS6 in HIV-infected pregnant women. This study will enroll pregnant women with and without HIV to receive GBS6 or Placebo in order to provide an expanded safety and immunogenicity data set (for both pregnant women and their infants) and to support progression of the development of this vaccine.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Maternal Participants

1. Age ≥ 18 to ≤ 40 years of age, inclusive at day of signing the ICF.
2. Pregnant at ≥ 27 0/7 to ≤35 6/7 gestation on the day of planned vaccination, verified by ultrasound scan (U/S).
3. Low risk, singleton pregnancy, as assessed by the study physician based on ultra-sound scan and previous obstetric history.
4. Documented negative HBV surface antigen, HCV antibody, and syphilis tests at screening.
5. Documented HIV test during pregnancy undertaken as per the national guidelines.
6. If HIV infected pregnant women, stable on ART for at least 3 months prior to study start
7. Determined by medical history, physical examination, screening laboratory assessment, and clinical judgment to be appropriate for inclusion in the study.
8. Receiving prenatal standard of care including HIV care if applicable at the clin-ics/physician offices/hospital network affiliated with the clinical study site.
9. Willing to give birth at Kawempe Specialised National Referral Hospital, or Kisenyi Health center IV, Uganda.
10. Willing and able to participate for the duration of the study visits and follow-up until 12-months post-delivery.
11. Willing and able to be contacted by telephone for the full duration of the study, and to give informed consent for their infant participant to participate in the study.

Inclusion criteria for Infants Inclusion criteria for Infants

1. Parent(s) willing and able to comply with scheduled visits, investigational plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Exclusion criteria for Maternal Participants

Any of the following:

1. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Pfizer employees, including their family members, directly involved in the conduct of the study.
2. Participants whose unborn baby have been fathered by investigational site staff members directly involved in the conduct of the study or their family members, site staff members otherwise supervised by the investigator, or Pfizer employees directly involved in the conduct of the study.
3. Participation in other studies involving investigational drug(s), vaccines, or medical devices within 28 days prior to study entry and/or during study participation.
4. Previous vaccination with any licensed or investigational GBS vaccine.
5. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the investigational product.
6. History of microbiologically proven invasive disease caused by GBS, or history of an infant with GBS disease.
7. Current alcohol abuse or illicit drug use.
8. Body mass index (BMI) of ≥40 kg/m2 at the time of the screening visit.
9. Clinical history of primary genital herpes simplex virus (HSV) infection during the current pregnancy.
10. A prior history of or current pregnancy complications or abnormalities that will increase the risk associated with the participant's participation in, and completion of, the study, including but not limited to the following (refer to the SRM) for further details):

    1. Gestational hypertension or preeclampsia eclampsia
    2. Placental abnormality
    3. Polyhydramnios or oligohydramnios
    4. Significant bleeding or blood clotting disorder
    5. Gestational diabetes
    6. Any signs of premature labour with the current pregnancy
11. Prior late stillbirth (defined as loss of pregnancy at any time after 28 weeks gestation) or neonatal death (defined as death of an infant within the first 28 days of life), prior low birth weight baby (defined as infant <2500 g) or premature delivery (defined as delivery before 37 0/7 weeks gestation), prior history of at least 3 miscarriages, prior pregnancies numbering greater than 5, or previous infant with a known or suspected genetic disorder or major congenital anomaly
12. Confirmed GBS bacteriuria during the current pregnancy
13. Major illness of the mother (outside of HIV serostatus) or conditions of the foetus that, in the investigator's judgment, will substantially increase the risk associated with the participant's participation in, and completion of, the study or could preclude the evaluation of the participant's response, including but not limited to the following (refer to the SRM) for further details):

    g. hypertension requiring treatment h. heart disease i. lung disease j. neurological disorders including a history of epilepsy or recurrent afebrile seizures k. kidney disease l. liver disease m. haematological disorders (including sickle cell disease) n. severe anaemia (less than 7.0g/dL) o. significant bleeding or blood clotting disorder p. endocrine disorders including known diabetes mellitus
14. Participants with known or suspected immunodeficiency (outside of HIV positive sero-status).
15. Participants who receive treatment with immunosuppressive therapy including cytotoxic agents or systemic corticosteroids, e.g., for cancer or an autoimmune disease, or planned receipt through the postvaccination blood draw. Inhaled/nebulised, intra articular, intra-bursal, or topical (skin or eyes) corticosteroids are permitted.
16. Receipt of blood/plasma products or immunoglobulin, from 60 days before investigational product administration, or planned receipt through delivery.
17. Known to be Rhesus Negative
18. Psychiatric condition including recent (within the last year) or active suicidal ideation or behaviour or laboratory abnormalities that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
19. Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalised involuntarily.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary mother outcome 1 | 7 days following administration of IMP
  1. Percentage Occurrence of solicited local reactions within 7 days following administration of investigational product (pain at the injection site, redness, and swelling).
Primary mother outcome 2 | 7 days following administration of IMP
  2. Percentage Occurrence of solicited systemic events within 7 days following administration of investigational product (fever, nausea/vomiting, diarrhoea, headache, fatigue/tiredness, muscle pain, and joint pain).
Primary mother outcome 3 | Through 1 month following administration of IMP
  3. Percentage Occurrence of solicited and unsolicited adverse events through 1 month after administration of investigational product.
Primary mother outcome 4 | Visit 1 through 12 months post-delivery
  4. Number Occurrence of SAEs, MAEs, and obstetric complications (peripartum, intrapartum, and postpartum) throughout the study (Visit 1 through the 12 month postdelivery study visit) and any unsolicited events leading to study withdrawal.
Primary Infant outcome 1 | Birth to 6 weeks of age
  1. Number Occurrence of unsolicited adverse events from birth to 6 weeks of age
Primary Infant outcome 2 | Through 12 months of age
  2. Number Occurrence of SAEs, AEs of special interest (major congenital anomalies, developmental delay, and suspected or confirmed GBS infection), and MAEs through 12 months of age and any unsolicited events leading to study withdrawal.

SECONDARY OUTCOMES:
Secondary mother Outcome 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV positive and HIV negative women | Baseline
  1. Geometric mean concentration GBS serotype specific IgG antibody titres measured at baseline in HIV positive and HIV negative women.
Secondary mother Outcome 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV positive and HIV negative women | 2 weeks after vaccination
  1. Geometric mean concentration GBS serotype specific IgG antibody titres measured at 2 weeks after vaccination in HIV positive and HIV negative women.
Secondary mother Outcome 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV positive and HIV negative women | 1 month after vaccination
  1. Geometric mean concentration GBS serotype specific IgG antibody titres measured at 1 month after vaccination in HIV positive and HIV negative women.
Secondary mother Outcome 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV positive and HIV negative women | Delivery
  1. Geometric mean concentration GBS serotype specific IgG antibody titres measured at delivery in HIV positive and HIV negative women.
Secondary mother Outcome 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV positive and HIV negative women | 6 weeks after delivery
  1. Geometric mean concentration GBS serotype specific IgG antibody titres measured at 6 weeks after delivery in HIV positive and HIV negative women.
Secondary Mother Objective 2 - Geometric mean concentration GBS serotype specific IgG titres in HIV positive and HIV negative women | Baseline
  2. Geometric mean concentration GBS serotype specific IgG titres measured at baseline in HIV positive and HIV negative women.
Secondary Mother Objective 2 - Geometric mean concentration GBS serotype specific IgG titres in HIV positive and HIV negative wome | Delivery
  2. Geometric mean concentration GBS serotype specific IgG titres measured at delivery in HIV positive and HIV negative women.
Secondary infant Objective 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV-exposed and unexposed infant participants | Birth
  1. Geometric mean concentration GBS serotype specific IgG antibody titres in HIV-exposed and unexposed infant participants measured at birth
Secondary infant Objective 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV-exposed and unexposed infant participants | 18 weeks
  1. Geometric mean concentration GBS serotype specific IgG antibody titres in HIV-exposed and unexposed infant participants measured at 18 weeks of life.
Secondary infant Objective 1 - Geometric mean concentration GBS serotype specific IgG antibody titres in HIV-exposed and unexposed infant participants | 12 months of life
  1. Geometric mean concentration GBS serotype specific IgG antibody titres in HIV-exposed and unexposed infant participants measured at 12 months of life.
Secondary infant Objective 2 - Geometric mean concentration GBS serotype specific IgG titres in HIV-exposed and unexposed infant participants | 18 weeks of life
  2. Geometric mean concentration GBS serotype specific IgG titres in HIV-exposed and unexposed infant participants measured at 18 weeks of life.
Secondary infant Objective 3 - Ratio Placental transfer ratio of GBS-specific antibodies in HIV-exposed and unexposed pregnancies. | Delivery
  3. Ratio Placental transfer ratio of GBS-specific antibodies in HIV-exposed and unexposed pregnancies.

OTHER OUTCOMES:
Mother Exploratory outcome 1 - Ratio Placental transfer ratio of GBS-specific antibodies in HIV-exposed and unexposed pregnancies. | Baseline through 12 months after delivery
  1. Fold increase in GBS serotype specific IgG antibody titres over baseline measured before vaccination through 12 months after delivery in HIV positive and HIV negative women.
Mother Exploratory outcome 2 - Percentage Serotype specific GBS positive vaginal and/or rectal culture(s) in HIV positive and HIV negative women. | Baseline
  2. Percentage Serotype specific GBS positive vaginal and/or rectal culture(s) before vaccination, at delivery, and 6 weeks after delivery in HIV positive and HIV negative women.
Mother Exploratory outcome 2 - Percentage Serotype specific GBS positive vaginal and/or rectal culture(s) in HIV positive and HIV negative women. | Delivery
  2. Percentage Serotype specific GBS positive vaginal and/or rectal culture(s) at delivery in HIV positive and HIV negative women.
Mother Exploratory outcome 2 - Percentage Serotype specific GBS positive vaginal and/or rectal culture(s) in HIV positive and HIV negative women. | 6 weeks after delivery
  2. Percentage Serotype specific GBS positive vaginal and/or rectal culture(s) at 6 weeks after delivery in HIV positive and HIV negative women.
Mother Exploratory outcome 3 - Concentration GBS serotype specific IgG and IgA antibody titres in breast milk following vaccination of women living with HIV and their unexposed counterparts | within 72 hours after delivery
  3. Concentration GBS serotype specific IgG and IgA antibody titres in breast milk following vaccination of women living with HIV and their unexposed counterparts in colostrum (within 72 hours of delivery)
Mother Exploratory outcome 3 - Concentration GBS serotype specific IgG and IgA antibody titres in breast milk following vaccination of women living with HIV and their unexposed counterparts | 6 weeks after delivery
  3. Concentration GBS serotype specific IgG and IgA antibody titres in breast milk following vaccination of women living with HIV and their unexposed counterparts in breast milk at 6 weeks after delivery.
Mother Exploratory outcome 3 - Concentration GBS serotype specific IgG and IgA antibody titres in breast milk following vaccination of women living with HIV and their unexposed counterparts | 18 weeks after delivery
  3. Concentration GBS serotype specific IgG and IgA antibody titres in breast milk following vaccination of women living with HIV and their unexposed counterparts in breast milk at 18 weeks after delivery.
Infant Exploratory outcome 1 - Concentration IgG antibody titres to vaccines included in the extended programme of vaccination administered to HIV-exposed and unexposed infant participants | 18 weeks of age
  Concentration IgG antibody titres to vaccines included in the extended programme of vaccination administered to HIV-exposed and unexposed infant participants as part of at 18 weeks of age
Infant Exploratory outcome 1 - Concentration IgG antibody titres to vaccines included in the extended programme of vaccination administered to HIV-exposed and unexposed infant participants | 12 months of age
  Concentration IgG antibody titres to vaccines included in the extended programme of vaccination administered to HIV-exposed and unexposed infant participants as part of at 12 months of age.
Infant Exploratory outcome 2 - Concentration Serotype specific GBS positive nasal/rectal cultures in infant participants | Delivery
  2. Concentration Serotype specific GBS positive nasal/rectal cultures at delivery in infant participants.
Infant Exploratory outcome 2 - Concentration Serotype specific GBS positive nasal/rectal cultures in infant participants | 6 weeks after delivery
  2. Concentration Serotype specific GBS positive nasal/rectal cultures at 6 weeks after delivery in infant participants.
Infant Exploratory outcome 2 - Concentration Serotype specific GBS positive nasal/rectal cultures in infant participants | 18 weeks after delivery
  2. Concentration Serotype specific GBS positive nasal/rectal cultures at 18 weeks after delivery in infant participants.
Infant Exploratory outcome 3 - Concentration GBS serotype specific IgG antibody titres measured from dried blood spots in infant participants. | At birth
  3. Concentration GBS serotype specific IgG antibody titres measured from dried blood spots in infant participants at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Musa sekikubo, Prof, Principal Investigator — Makerere University - John Hopkins University
Locations (1):
- Makerere University, John Hopkins University, Kawempe, Uganda

DOCUMENTS (1):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT05832502/Prot_001.pdf